CLINICAL TRIAL: NCT01160250
Title: A Single-Arm, Open-Label, Expanded Access Study of Vismodegib (GDC-0449) in Patients With Locally Advanced or Metastatic Basal Cell Carcinoma
Brief Title: A Study of Vismodegib (GDC-0449) in Patients With Locally Advanced or Metastatic Basal Cell Carcinoma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SHH4811g
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

INTERVENTIONS:
Drug: vismodegib (GDC-0449) — Oral repeating dose

SUMMARY:
This is an open-label, non-comparative, multicenter, expanded access study of Vismodegib (GDC-0449) in patients with locally advanced basal cell carcinoma (BCC) or metastatic BCC (mBCC) who are otherwise without satisfactory treatment options.

ELIGIBILITY:
Inclusion Criteria:

* For patients with mBCC, histologic confirmation of distant BCC metastasis
* For patients with locally advanced BCC, at least one histologically confirmed lesion 10 mm or more in diameter and written confirmation from a surgical specialist that the tumor is considered inoperable or that surgery is contraindicated
* For patients with locally advanced BCC, radiotherapy must have been previously administered for locally advanced BCC, unless radiotherapy is contraindicated or inappropriate. For patients whose locally advanced BCC has been irradiated, disease must have progressed after radiation.
* Patients with Gorlin syndrome may enroll in this study but must meet the criteria for locally advanced or metastatic disease listed above
* Patients with measurable and/or non-measurable disease (as defined by RECIST) are allowed
* Adequate organ function
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception, including one barrier method, during the study and for 12 months after discontinuation of Vismodegib (GDC-0449)
* For men with female partners of childbearing potential, agreement to use a latex condom, and to advise their female partner to use an additional method of contraception during the study and for 3 months after discontinuation of Vismodegib (GDC-0449)

Exclusion Criteria:

* Pregnancy or lactation
* Life expectancy < 12 weeks
* Concurrent non-protocol-specified anti-tumor therapy
* Completion of most recent anti-tumor therapy at least 21 days prior to initiation of treatment
* Uncontrolled medical illnesses such as infection requiring treatment with intravenous antibiotics
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or renders the patient at high risk from treatment complications
* Unwillingness to practice effective birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (10):
  - Scottsdale, Arizona
  - Los Angeles, California
  - Stanford, California
  - Ormond Beach, Florida
  - Detroit, Michigan
  - New York, New York
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas

REFERENCES:
- [Derived] Chang AL, Arron ST, Migden MR, Solomon JA, Yoo S, Day BM, McKenna EF, Sekulic A. Safety and efficacy of vismodegib in patients with basal cell carcinoma nevus syndrome: pooled analysis of two trials. Orphanet J Rare Dis. 2016 Sep 1;11(1):120. doi: 10.1186/s13023-016-0506-z. PMID 27581207